CLINICAL TRIAL: NCT01901081
Title: A Feasibility Study to Assess Safety and Functionality of Implantable Myoelectric Sensors for Upper Extremity Prosthetic Control in Transradial Amputees
Brief Title: Feasibility of Implantable Myoelectric Sensors to Control Upper Limb Prostheses
Acronym: IMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred E. Mann Foundation for Scientific Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP0015B
Record Dates: First submitted 2013-05-20; First posted 2013-07-17 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Amputation, Traumatic
Keywords: Implantable Myoelectric Sensor; IMES; transradial; amputation; myoelectric; prosthesis; prosthetic control
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prosthetic Training with IMES prosthesis (Experimental)
  Interventions: Device: IMES

INTERVENTIONS:
Device: IMES — Once subjects recover from surgical implantation of IMES (approximately two weeks), they will practice IMES control using a bench-top IMES trainer for approximately a month. As soon as the subject's custom-fit IMES Prosthesis is available, it will be fitted and programmed. Subjects will then begin six months of prosthetic training. Month 1 training entails sessions with an Occupational Therapists 4-5 times per week. Months 2-6 Training entail meeting with an Occupational Therapist twice a month. During training, subject will learn how to contract residual musculature in the amputated limb to control movements of an electromechanical wrist and hand. The therapeutic goal is to develop skills needed to perform Activities of Daily Living using the IMES prosthesis.
  After completing six months of training, subjects will be given the option to continue using their IMES Prosthesis for another sixteen months.
  Other Names: Myoelectric Prosthetic Training

SUMMARY:
This study will evaluate the feasibility of using implanted myoelectric sensors (IMES) to control an electromechanical prosthetic wrist and hand.

DETAILED DESCRIPTION:
The study assesses the feasibility of an advanced prosthesis control system aimed at development of a more intuitive and functional prosthetic device. Tiny (2.5 mm by 16 mm) Implantable Myoelectric Sensors (IMES) will be implanted into the residual forearm muscles of three transradial amputee subjects. These devices wirelessly transmit electrical muscle signals to an electromechanical prosthetic wrist and hand.

Following a two-week recovery from implantation of six to eight IMES into residual forearm muscles, subjects will initiate seven months of training. Subjects first train for approximately a month using a bench-top IMES system. When they receive their custom-fit IMES Prosthesis (including electromechanical wrist and hand) subjects initiate six months of additional training. Subjects will then be given the option to use the IMES Prosthesis for another sixteen months. The usability and functionality of the prosthetic system will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a health care beneficiary at the Walter Reed National Military Medical Center.
2. Patient has transradial amputation with one-third or greater residual forearm length as determined by the contralateral side.
3. Patient's residual forearm anatomy (based on number and size of residual muscles) will support the implantation and control of at least six IMES (in the opinion of the Investigator). This criterion will be verified during a study-specific screening test.
4. Patient is age 18 or above.
5. Patient can speak and comprehend English.
6. Patient is willing and capable of providing informed consent.
7. Patient has undergone amputee rehabilitation, including being trained to wear and use a body-powered and myoelectric prosthesis.
8. Patient reports wearing an upper limb prosthesis at least two hours per day.
9. Unilateral amputation with preserved function of the non-amputated arm; preserved function is investigator opinion as to whether the patient:

   * has the ability to independently don and doff a prosthesis,
   * has enough dexterity in the non-amputated arm to attach and detach the Prosthetic Control Interface (PCI) cable and operate the PCI power switch,
   * has the dexterity to remove and replace the PCI battery.
10. Patient is willing and capable of having EMG needles inserted into the forearm.
11. In the opinion of the Investigator, patient is cognitively capable of operating an IMES Prosthesis.
12. Patient is willing to comply with a wearing schedule for the investigational device.
13. Patient is willing and capable of travelling to the investigational site for study visits outlined in this protocol.

Exclusion Criteria:

1. Patient is less than three months from amputation surgery or major injury of the target residual limb.
2. Patient has major injury proximal to the level of amputation.
3. In the opinion of the Investigator, patient is prone to skin breakdown in the target residual limb.
4. Known nerve transection or palsy that may cause de-innervation of muscles in the target residual limb.
5. Known genetic neuromuscular disorder (e.g. multiple sclerosis, myasthenia gravis, muscular dystrophy).
6. Patient has a bleeding or clotting disorder.
7. Bilateral upper extremity amputation.
8. Patient has a major psychological disorder such as poorly controlled PTSD, schizophrenia, or paranoia such that cooperative status is inconsistent.
9. Patient has an active implant (e.g. pacemaker, implanted cardiac defibrillator [ICD], neurostimulator, drug infusion device).
10. Patients having any metal fragments or metal implants (e.g. orthopedic hardware) located within the residual forearm are excluded. The absence of metal shall be confirmed by an x-ray of the entire affected arm.
11. Patients having metal in the affected upper arm will be considered on a case-by-case basis. An x-ray of the entire affected arm shall be provided to the Sponsor who will assess potential interaction of the metal with the Coil's magnetic field.
12. Patient has a history of adverse reactions to anesthetic agents.
13. Patient has recently or is currently participating in research that may influence response to either study intervention, or be harmful to the subject in any way.
14. A female patient who is pregnant, nursing, or planning to become pregnant during the course of the study.
15. In the opinion of the Investigator, the subject is not a suitable candidate for the study, for any reason such as residual limb infection, significant pain, significant proximal nerve injury or soft tissue damage, significant scarring, or poor health of the skin envelope.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Device-Related Serious Adverse Events | Information collected over the course of 2 years following implant of IMES
  Tabulation of Device-Related Serious Adverse Events during the course of the study.
Change in Accuracy Test score | test conducted nine times: upon receipt and programming of custom-fit IMES prosthesis; once per month for six months of training; 1 year following implant; and 2 years following implant
  The Accuracy Test requires subjects to execute a series of different hand movements using the IMES to control an electromechanical wrist and hand. Movements are chosen to demonstrate both independent and simultaneous control over the six different movements offered by the prosthesis: hand open/close, thumb adduct/abduct, wrist supinate/pronate. An occupation therapist will score the subject on each movement as follows: 0 = no movement observed; 1 = the intended movement was not observed, but unintended movements were observed; 2 = the intended movement was observed, in addition to unintended movements; 3 = the intended movement was observed. The change in Accuracy Scores across the nine tests completed will be presented.
  During the Accuracy Test, Electromyographic(EMG) signals transmitted by the IMES will be recorded. A video camera will record the movements of the prosthesis so that this output may be associated with the input IMES signals.

SECONDARY OUTCOMES:
Change in Southampton Hand Assessment Procedure (SHAP) test score | test conducted nine times: upon receipt and programming of custom-fit IMES prosthesis; once per month for six months of training; 1 year following implant; and 2 years following implant
  The test entails a series of self-timed tasks (the participant starting and stopping the timer with the hand under test), which are divided into two sections: picking and placing eight different shaped objects and performing fourteen Activities of Daily Living (ADL). The objects are shaped to encourage the use of six standard prehensile patterns (spherical, tripod, power, lateral, tip, extension) and come in two different weights to test the participant's ability to form more powerful grips. The fourteen simulated ADLs include cutting, pouring, lifting and transferring loads. Subjects will perform the SHAP test using the IMES to control an electromechanical wrist and hand. Each task is scored based on the amount of time to complete. The change in SHAP scores across the nine tests completed will be presented.
Change in Assessment of Capacity for Myoelectric Control (ACMC) test score | test conducted nine times: upon receipt and programming of custom-fit IMES prosthesis; once per month for six months of training; 1 year following implant; and 2 years following implant
  The ACMC is administered and scored based on observations of the subject as he or she is performing an everyday task using the IMES to control an electromechanical wrist and hand. Tasks will be chosen from a selection of six that include: packing a suitcase, sorting mail, mixing a ready-to-eat product, repotting a plant, assembling a ready-made project, and setting a table. During the assessment, subjects are encouraged to accomplish the task spontaneously in their usual way. The occupational therapist assesses capacity for control of the prosthesis by rating the performances on 22 items representing different aspects of control that are classified as gripping, holding, releasing, and coordinating between hands. Each subject's performance is rated with scores ranging from 0 to 3, where 0 = not capable, 1 = sometimes capable, capacity not established, 2 = capable on request, and 3 = spontaneously capable. The change in ACMC Scores across the nine tests completed will be presented.
Change in Box and Block Test (BBT) score | test conducted nine times: upon receipt and programming of custom-fit IMES prosthesis; once per month for six months of training; 1 year following implant; and 2 years following implant
  The BBT measures unilateral gross manual dexterity. The BBT is composed of a wooden box divided in two compartments and 150 blocks. The subject is asked to move as many blocks as possible from one compartment of a box to another, within 60 seconds. The task is to be performed using the IMES to control an electromechanical wrist and hand. The change in BBT Score across the nine tests completed will be presented.
IMES Satisfaction Questionnaire | completed after six months of training following upon receipt and programming of custom-fit IMES prosthesis
  Subjects will be asked to complete a questionnaire in which they rate and describe their satisfaction with different aspects of the IMES Prosthesis.

OTHER OUTCOMES:
Device Malfunctions | Information collected over the course of 2 years following implant of IMES
  A frequency table will be provided to summarize the type and number of all Device Malfunctions during the course of the study.
IMES System Usage | information collected over the course of 6 months following upon receipt and programming of custom-fit IMES prosthesis
  The number of hours and types of usage will be summarized for each subject
Programming Requirements | Information collected over the course of 2 years following implant of IMES
  The number of hours and sessions required to program the IMES Prosthesis for each subject over the course of their participation in the study will be presented in a table.
  IMES parameter settings (control signal and gain) recorded at each Programming Visit for all implanted IMES will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Pasquina, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States